CLINICAL TRIAL: NCT06293482
Title: A Pivotal, Prospective, Open-label, Multi-center Study of Safety and Effectiveness of Cochlear Implantation in an Expanded Population of Adults With Bilateral Sensorineural Hearing Loss
Brief Title: Safety and Effectiveness of Cochlear Implantation in an Expanded Adult Population
Acronym: ACE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: NAMSA (Other); LWB Consulting (Unknown); Althea Anagnostopoulos Harrington (Unknown); MV Clinical Research, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM5850
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-03

CONDITIONS: Hearing Loss, Sensorineural; Hearing Loss, Bilateral
Keywords: Cochlear implant; Sensorineural hearing loss; Safety; Efficacy
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss, Bilateral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Cochlear™ Nucleus® System (Experimental): Participants will be implanted with a commercially approved Cochlear™ Nucleus® implant.
  Interventions: Device: Cochlear™ Nucleus® System

INTERVENTIONS:
Device: Cochlear™ Nucleus® System — The Cochlear™ Nucleus ® System is a commercially available system intended for restoration of hearing sensation through electrical stimulation of the auditory nerve in adult patients with bilateral symmetrical sensorineural hearing loss.

SUMMARY:
This study aims to evaluate the safety and efficacy of cochlear implantation for adults with bilateral sensorineural hearing loss who currently do not meet the FDA-approved indications for cochlear implantation. Following cochlear implantation, participants will complete speech perception assessments and questionnaires over the course of seven visits.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18 or older at the time of consent
* Meets the following audiometric criteria for the ear to be implanted: clinically established sensorineural hearing loss (SNHL) defined by a four frequency pure tone average (PTA) at 500, 1000, 2000, & 4000 Hz of: ≥60 dB HL and compromised functional hearing in the aided condition defined as <50% correct on a word recognition test
* Meets the following audiometric criteria for the non-implanted contralateral ear: clinically established SNHL defined by a four frequency PTA at 500, 1000, 2000, & 4000 Hz of >30 dB HL
* Candidate is a fluent speaker in the language used to assess speech perception performance as determined by the investigator.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Meets current indications on audiometric thresholds for traditional adult CI candidates (i.e., bilateral moderate to profound hearing loss in the low frequencies and profound [≥ 90 dB HL] hearing loss in the mid to high speech frequencies)
* Absence of cochlea development or a cochlear nerve
* Presence of active middle ear infection in the ear to be implanted
* Tympanic membrane perforation in the presence of active middle ear disease in the ear to be implanted
* Medical or psychological conditions that contraindicate general anaesthesia, surgery, or participation in the clinical investigation.
* Existing contralateral cochlear implant or medical plan to implant a contralateral cochlear implant during the clinical investigation.
* Pregnant or breastfeeding women. Women who plan to become pregnant during the course of the clinical investigation.
* Unrealistic expectations on the part of the participant, regarding the possible benefits, risks, and limitations that are inherent to the surgical procedure(s) and prosthetic devices as determined by the investigator.
* Additional disabilities that may affect the participant's participation of safety during the clinical investigation.
* Unable or unwilling to comply with all of the requirements of the clinical investigation as determined by the investigator.
* Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
* Employees of Cochlear.
* Current participation, or participation in another interventional clinical study/trial in the past 30 days, involving an investigational drug or device (unless the other investigation was/is a Cochlear sponsored investigation and determined by the investigator or Sponsor to not impact this investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Number of device and procedure-related adverse events and serious adverse events | 6-months post-activation
  Events will be summarized by type, frequency, and severity.
Mean change on aided word recognition in the unilateral CI alone listening condition at 6 months post-activation compared to pre-operative baseline in the unilateral aided listening condition for the ear to be implanted | Pre-operative baseline, 6 months post-activation
  The CNC word recognition test (for English speakers) and Spanish Bisyllabic word test (for Spanish speakers) will be administered in quiet at a level equal to 60dBA in the sound field. The tests will be scored as total number of words correct, which will be expressed as a percentage correct for this study.
Mean change on AzBio sentences in noise at 6 months post-activation in the everyday listening condition compared to pre-operative performance in the everyday listening condition | Pre-operative baseline, 6 months post-activation
  The AzBio sentence test (for English speakers) and the Spanish AzBio sentence test (for Spanish speakers) will be utilised. These are validated tests to assess the open-set sentence recognition in quiet or in the presence of competing noise. For this study, the target sentences will be presented at a fixed level of 65dBA starting at a +10 dB signal-to-noise ratio using multi-talker babble as the competing signal. Each word in the sentence counts towards the overall score, which will be expressed as a percent correct for this study.

SECONDARY OUTCOMES:
Number of device and procedure related adverse events and serious adverse events | 36-Months post-activation
  Events will be summarized by type, frequency, and severity.
Proportion of participants who demonstrate a change score of +1 or greater on the Speech, Spatial and Qualities of Hearing Scale (SSQ12) at 6-months post-activation compared to preoperative baseline | Pre-operative baseline, 6 months post-activation
  The SSQ12 is a self-administered questionnaire designed to measure auditory disability across three categories: speech perception, spatial hearing, and qualities of hearing. Respondents rate their perceived ability or experience for each scenario questioned on a 'ruler' (horizontal line) that is numbered, left to right, from '0' corresponding to no ability, to '10,' corresponding to complete ability. Higher scores represent greater ability.
Mean change on the Tinnitus Handicap Inventory (THI) score at 6-months post-activation compared to preoperative baseline will exceed a 7-point improvement | Pre-operative baseline, 6 months post-activation
  The THI is a 25-item self-assessment questionnaire used to assess the impact of tinnitus on a patient's quality of life. Items are grouped into functional, emotional, and catastrophic domains. A "yes" response is scored with 4 points; "sometimes" with 2 points; and "no" with zero points. Scores for the total scale range from 0 to 100 points, with higher scores representing greater perceived handicap.
Mean change on aided word recognition in the unilateral CI alone listening condition at 3 months post activation compared to pre-operative baseline in the unilateral aided listening condition for the ear to be implanted | Pre-operative baseline, 3 months post-activation
  The CNC word recognition test (for English speakers) and Spanish Bisyllabic word test (for Spanish speakers) will be administered in quiet at a level equal to 60dBA in the sound field. The tests will be scored as total number of words correct, which will be expressed as a percentage correct for this study.
Mean change on AzBio sentences in noise at 3 months post-activation in the everyday listening condition compared to pre-operative performance in the everyday listening condition | Pre-operative baseline, 3 months post-activation
  The AzBio sentence test (for English speakers) and the Spanish AzBio sentence test (for Spanish speakers) will be utilised. These are validated tests to assess the open-set sentence recognition in quiet or in the presence of competing noise. For this study, the target sentences will be presented at a fixed level of 65dBA starting at a +10 dB signal-to-noise ratio using multi-talker babble as the competing signal. Each word in the sentence counts towards the overall score, which will be expressed as a percent correct for this study.
Percentage correct on aided word recognition in the unilateral condition in the implanted ear in the post-operative everyday listening condition | 6 months post-activation
  This will be evaluated for those participants who have a LFPTA (125-500 Hz) <80 dB HL versus those participants who have a LFPTA (125-500 Hz) ≥ 80 dB HL.
Percentage correct on AzBio sentences in noise in the post-operative everyday listening condition | 6 months post-activation
  This will be evaluated for those participants who have a LFPTA (125-500 Hz) <80 dB HL versus those participants who have a LFPTA (125-500 Hz) ≥ 80 dB HL.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Centre for Neurosciences, Tucson, Arizona
  - Pacific Neuroscience Institute, Santa Monica, California
  - University of Miami, Coral Gables, Florida
  - Indiana University, Indianapolis, Indiana
  - Midwest Ear Institute, Kansas City, Missouri
  - New York University, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania Hospitals, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Cochlear do not have an approved platform for public sharing of IPD collected in this study. Data may be provided to individual researchers on request.